CLINICAL TRIAL: NCT03379350
Title: The Impacts of Intermittent Chest Tube Clamping on Chest Tube Drainage Duration and Postoperative Hospital Stay After Lung Cancer Surgery: A Prospective Study
Brief Title: The Impacts of Intermittent Chest Tube Clamping on Chest Tube Drainage Duration and Postoperative Hospital Stay After Lung Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wu Nan (Other)
Responsible Party: Sponsor-Investigator, Wu Nan, Assistant of hospital director, Peking University Cancer Hospital & Institute
Organization: Peking University Cancer Hospital & Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10574
Record Dates: First submitted 2017-09-30; First posted 2017-12-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Management of Lung Cancer Patients
Keywords: lung cancer; surgery; chest tube clamping; duration of chest tube drainage; postoperative stay
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- clamping group (Experimental): Clamping group are managed with clamping protocol after 3pm on the postoperative day as follow: the chest tube will be clamped, and the nurses will check the patient every 6 h. If the patient has no problems with compliance, the clamp will be removed for half an hour in the morning to record the drainage volume every 24 h.
  Interventions: Procedure: clamping group
- control group (No Intervention): Patients in control group are managed with gravity drainage (water seal only, without suction) all the time after operation.

INTERVENTIONS:
Procedure: clamping group — Clamping group are managed with clamping protocol after 3pm on the postoperative day as follow: the chest tube will be clamped, and the nurses will check the patient every 6 h. If the patient has no problems with compliance, the clamp will be removed for half an hour in the morning to record the drainage volume every 24 h.
  Arms: clamping group

SUMMARY:
All patients undergo lateral thoracotomy or video-assisted thoracoscopic surgery (VATS) and are operated on by the same thoracic surgical team. All patients are managed with gravity drainage (water seal only, without suction) on the day of operation. Eligible patients are randomized to control group or clamping group at a 1:1 ratio before 3pm on the postoperative day. Patients in control group and those in clamping group are managed with different protocols after 3pm on the postoperative day.

DETAILED DESCRIPTION:
All patients undergo lateral thoracotomy or video-assisted thoracoscopic surgery (VATS) and are operated on by the same thoracic surgical team. At the end of operation, the lung parenchyma is submerged in sterile saline to test for air leakage, and a single 24-Fr chest tube is placed in each patient. All patients are managed with gravity drainage (water seal only, without suction) on the day of operation.

Once a radiograph is confirmed re-expansion of the lung on the morning of the first postoperative day and no air leak is detected, the patient is a candidate for inclusion in the trial. Eligible patients are randomized to control group or clamping group before 3pm on the postoperative day.

Patients in control group are managed with gravity drainage unchangeably, while patients in clamping group are managed with clamping protocol after 3pm on the postoperative day as follow: the chest tube will be clamped, and the nurses will check the patient every 6 h. If the patient has no problems with compliance, the clamp will be removed for half an hour in the morning to record the drainage volume every 24 h. If patients develops intolerable abnormal symptoms, such as dyspnea, pneumothorax, and severe subcutaneous emphysema after chest tube clamping, the clamp will be removed for 30 min and be reapplied after the symptoms have been resolved. Such patients will be placed under more rigorous surveillance after re-clamping, which requires the medical staff to check on the patients every 2-4 hours in order to promptly detect abnormal symptoms. If abnormal symptoms occur frequently, this clamping protocol will be continued until another radiograph excluded the presence of pneumothorax.

The daily output of pleural fluid was recorded. The criteria for chest tube removal were as follows: (a) drainage volume≤250 mL in 24 h, (b) absence of air leakage and intrathoracic hemorrhage, and (c) absence of signs of purulent pleural effusion and atelectasis.

ELIGIBILITY:
Inclusion Criteria:

Pathological diagnosis of lung cancer Treated with lobectomy and systematic mediastinal lymph node dissection/ systematic sampling Managed with gravity drainage (water seal only, without suction) Re-expansion of the lung confirmed on the morning of the first postoperative day

Exclusion Criteria:

Thoracic cavity infection Prolonged air leakage Reoperation due to chylothorax Atelectasis Liver cirrhosis Renal insufficiency Wound infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-05-28 (Actual)

PRIMARY OUTCOMES:
chest tube drainage duration | From date of operation until the date of chest tube removal, assessed up to 10 days
  time from operation day to the day of chest tube removal

SECONDARY OUTCOMES:
postoperative hospital stay | From date of operation until the date of hospital discharge, assessed up to 2 weeks
  time from opertion day to the day of hospital discharge

OTHER OUTCOMES:
decrease of hemoglobin level | postoperative day 1, before hosptital discharge and 1 month after the operation
  the decrease of hemoglobin on the first postoperative day and before discharge and a month after surgery
decrease of serum albumin level | postoperative day 1, before hosptital discharge and 1 month after the operation
  the decrease of serum albumin on the first postoperative day and before discharge and a month after surgery
pleural effusion thickness | observed through CT scan 1 month after the operation
  pleural effusion thickness showed on the CT scan a month after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Wang Y, Pei Y, Lv C, Wang Y, Wang J, Zhao D, Li X, Yang Y, Kim AW, Toker A, Yan S, Wu N. Intermittent chest tube clamping decreases chest tube duration time and drainage volume after lung cancer surgery in patients without air leak: an open-label, randomized controlled trial. Transl Lung Cancer Res. 2022 Mar;11(3):357-365. doi: 10.21037/tlcr-22-150. PMID 35399576